CLINICAL TRIAL: NCT05382442
Title: A Phase II Study of AK112 With or Without AK117 for Patients With Metastatic Colorectal Cancer
Brief Title: A Study of AK112 With or Without AK117 in Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-206
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (11):
- Part 1_Chemotherapy Regimen Selection Stage Group A(AK112+AK117+XELOX) (Experimental): AK112+AK117+XELOX
  AK112 and AK117 and XELOX(Oxaliplatin 130 mg/sqm iv day 1, Capecitabine via oral, the total daily dose was 2000mg/sqm, day1-14)
  If no progression occurs during AK112 plus AK117 plus XELOX, patients will receive maintenance capecitabine plus AK112 plus AK117 at the same dose used at the last cycle of the induction treatment. Capecitabine plus AK112 plus AK117 will be repeated every 3 weeks until disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: AK112; Drug: AK117; Drug: Oxaliplatin; Drug: Capecitabine
- Part 1_Chemotherapy Regimen Selection Stage Group B(AK112+AK117+FOLFOXIRI) (Experimental): AK112+AK117+FOLFOXIRI
  AK112 and AK117 and FOLFOXIRI(Irinotecan 150-165 mg/sqm iv day 1, Oxaliplatin 85 mg/sqm iv day 1, Leucovorin(LV) 400 mg/sqm iv day 1, 5-fluorouracil(5-FU) 2400-2800 mg/sqm 46-48 hours continuous infusion, starting on day 1)
  If no progression occurs during AK112 plus AK117 plus FOLFOXIRI, patients will receive maintenance 5-FU/LV plus AK112 plus AK117 at the same dose used at the last cycle of the induction treatment. 5-FU/LV plus AK112 plus AK117 will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: AK112; Drug: AK117; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-fluorouracil
- Part 1_Expansion Stage Group A(AK112 DS1+Chemotherapy) (Experimental): AK112 (Dose1) +Chemotherapy(Decided by Chemotherapy Regimen Selection Stage)
  AK112 and XELOX or FOLFOXIRI(the same dosage, frequency and duration with Chemotherapy Regimen Selection Stage)
  Interventions: Drug: AK112; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-fluorouracil
- Part 1_Expansion Stage Group B(AK112 DS1+AK117 DS1+Chemotherapy) (Experimental): AK112 (Dose1) +AK117 (Dose1) +Chemotherapy(Decided by Chemotherapy Regimen Selection Stage)
  AK112 and AK117 and XELOX or FOLFOXIRI(the same dosage, frequency and duration with Chemotherapy Regimen Selection Stage)
  Interventions: Drug: AK112; Drug: AK117; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-fluorouracil
- Part 1_Expansion Stage Group C (AK112 DS2+Chemotherapy) (Experimental): AK112 (Dose2)+Chemotherapy(Decided by Chemotherapy Regimen Selection Stage). AK112 and XELOX or FOLFOXIRI(the same dosage, frequency and duration with Chemotherapy Regimen Selection Stage).
  Interventions: Drug: AK112; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-fluorouracil
- Part 1_Expansion Stage Group D (AK112 DS2 +AK117 DS2 +Chemotherapy) (Experimental): AK112(Dose2) + AK117(Dose2)+Chemotherapy(Decided by Chemotherapy Regimen Selection Stage) AK112 and AK117 and XELOX or FOLFOXIRI(the same dosage, frequency and duration with Chemotherapy Regimen Selection Stage)
  Interventions: Drug: AK112; Drug: AK117; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-fluorouracil
- Part 1_Expansion Stage Group E (AK112 DS2+AK117 DS1+Chemotherapy) (Experimental): AK112(Dose2)+AK117(Dose1)+Chemotherapy(Decided by Chemotherapy Regimen Selection Stage) AK112 and AK117 and XELOX or FOLFOXIRI(the same dosage, frequency and duration with Chemotherapy Regimen Selection Stage)
  Interventions: Drug: AK112; Drug: AK117; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-fluorouracil
- Part 1_Extension Stage Group F (AK112 DS1 + mFOLFOX6) (Experimental): AK112 (Dose1) +mFOLFOX6 ( Oxaliplatin 85 mg/sqm IV day 1, Leucovorin 400 mg/sqm IV day 1, 5-fluorouracil(5-FU) 2400 mg/sqm 46-48 hours continuous infusion, starting on day 1).
  If no progression occurs during AK112 plus mFOLFOX6, patients will receive maintenance 5- FU/LV plus AK112 at the same dose used at the last cycle of the induction treatment. 5-FU/LV plus AK112 will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: AK112; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-fluorouracil
- Part 1_Extension Stage Group G (AK112 DS2+mFOLFOX6) (Experimental): AK112 (Dose2) +mFOLFOX6 ( Oxaliplatin 85 mg/sqm IV day 1, Leucovorin 400 mg/sqm IV day 1, 5-fluorouracil(5-FU) 2400 mg/sqm 46-48 hours continuous infusion, starting on day 1)
  If no progression occurs during AK112 plus mFOLFOX6, patients will receive maintenance 5- FU/LV plus AK112 at the same dose used at the last cycle of the induction treatment. 5-FU/LV plus AK112 will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: AK112; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-fluorouracil
- Part 2 cohort 1(AK112) (Experimental): Subjects receive AK112 until disease progression or unacceptable toxicity AK112 (until disease progression, unacceptable toxicity or patient's refusal)
  Interventions: Drug: AK112
- Part 2 cohort 2(AK112+AK117) (Experimental): Subjects receive AK117 and AK112 until disease progression or unacceptable toxicity AK112 and AK117 ( until disease progression, unacceptable toxicity or patient's refusal)
  Interventions: Drug: AK112; Drug: AK117

INTERVENTIONS:
Drug: AK112 — AK112 via intravenous (IV) infusion until disease progression or unacceptable toxicity
Drug: AK117 — AK117 via intravenous (IV) infusion until disease progression or unacceptable toxicity
  Arms: Part 1_Chemotherapy Regimen Selection Stage Group A(AK112+AK117+XELOX); Part 1_Chemotherapy Regimen Selection Stage Group B(AK112+AK117+FOLFOXIRI); Part 1_Expansion Stage Group B(AK112 DS1+AK117 DS1+Chemotherapy); Part 1_Expansion Stage Group D (AK112 DS2 +AK117 DS2 +Chemotherapy); Part 1_Expansion Stage Group E (AK112 DS2+AK117 DS1+Chemotherapy); Part 2 cohort 2(AK112+AK117)
Drug: Oxaliplatin — Oxaliplatin via IV infusion
  Arms: Part 1_Chemotherapy Regimen Selection Stage Group A(AK112+AK117+XELOX); Part 1_Chemotherapy Regimen Selection Stage Group B(AK112+AK117+FOLFOXIRI); Part 1_Expansion Stage Group A(AK112 DS1+Chemotherapy); Part 1_Expansion Stage Group B(AK112 DS1+AK117 DS1+Chemotherapy); Part 1_Expansion Stage Group C (AK112 DS2+Chemotherapy); Part 1_Expansion Stage Group D (AK112 DS2 +AK117 DS2 +Chemotherapy); Part 1_Expansion Stage Group E (AK112 DS2+AK117 DS1+Chemotherapy); Part 1_Extension Stage Group F (AK112 DS1 + mFOLFOX6); Part 1_Extension Stage Group G (AK112 DS2+mFOLFOX6)
Drug: Capecitabine — Capecitabine via oral,The total daily dose was 2000mg/sqm, Each cycle was administered for 2 consecutive weeks, followed by a week of rest, with a treatment cycle every 21 days
  Arms: Part 1_Chemotherapy Regimen Selection Stage Group A(AK112+AK117+XELOX); Part 1_Expansion Stage Group A(AK112 DS1+Chemotherapy); Part 1_Expansion Stage Group B(AK112 DS1+AK117 DS1+Chemotherapy); Part 1_Expansion Stage Group C (AK112 DS2+Chemotherapy); Part 1_Expansion Stage Group D (AK112 DS2 +AK117 DS2 +Chemotherapy); Part 1_Expansion Stage Group E (AK112 DS2+AK117 DS1+Chemotherapy)
Drug: Irinotecan — Irinotecan via IV infusion
  Arms: Part 1_Chemotherapy Regimen Selection Stage Group B(AK112+AK117+FOLFOXIRI); Part 1_Expansion Stage Group A(AK112 DS1+Chemotherapy); Part 1_Expansion Stage Group B(AK112 DS1+AK117 DS1+Chemotherapy); Part 1_Expansion Stage Group C (AK112 DS2+Chemotherapy); Part 1_Expansion Stage Group D (AK112 DS2 +AK117 DS2 +Chemotherapy); Part 1_Expansion Stage Group E (AK112 DS2+AK117 DS1+Chemotherapy)
Drug: Leucovorin — Leucovorin via IV infusion
  Arms: Part 1_Chemotherapy Regimen Selection Stage Group B(AK112+AK117+FOLFOXIRI); Part 1_Expansion Stage Group A(AK112 DS1+Chemotherapy); Part 1_Expansion Stage Group B(AK112 DS1+AK117 DS1+Chemotherapy); Part 1_Expansion Stage Group C (AK112 DS2+Chemotherapy); Part 1_Expansion Stage Group D (AK112 DS2 +AK117 DS2 +Chemotherapy); Part 1_Expansion Stage Group E (AK112 DS2+AK117 DS1+Chemotherapy); Part 1_Extension Stage Group F (AK112 DS1 + mFOLFOX6); Part 1_Extension Stage Group G (AK112 DS2+mFOLFOX6)
Drug: 5-fluorouracil — 5-fluorouracil via IV infusion
  Arms: Part 1_Chemotherapy Regimen Selection Stage Group B(AK112+AK117+FOLFOXIRI); Part 1_Expansion Stage Group A(AK112 DS1+Chemotherapy); Part 1_Expansion Stage Group B(AK112 DS1+AK117 DS1+Chemotherapy); Part 1_Expansion Stage Group C (AK112 DS2+Chemotherapy); Part 1_Expansion Stage Group D (AK112 DS2 +AK117 DS2 +Chemotherapy); Part 1_Expansion Stage Group E (AK112 DS2+AK117 DS1+Chemotherapy); Part 1_Extension Stage Group F (AK112 DS1 + mFOLFOX6); Part 1_Extension Stage Group G (AK112 DS2+mFOLFOX6)

SUMMARY:
This trial is a Phase II study. The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of AK112 with or without AK117 in participants with metastatic colorectal cancer who are not suitable for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of colorectal adenocarcinoma
* Part1: Subjects who have not previously received any systemic antitumor therapy and who have previously received neoadjuvant or adjuvant therapy, the first detection of recurrence or metastasis should be ≥12 months after the last administration of neoadjuvant or adjuvant therapy
* Part2: Subjects who have previously received systemic therapy including fluorouracil, oxaliplatin, irinotecan, bevacizumab or anti-EGFR antibodies or could not tolerate or have contraindications to standard treatment
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Measurable disease as defined by RECIST v1.1
* Adequate hematologic and organ function

Exclusion Criteria:

* Known MSI-H(Microsatellite-Instability-High) or dMMR(Mismatch Repair-Deficient)
* Prior treatment with immunotherapy, including immune checkpoint inhibitors , immune checkpoint agonists, immune cell therapy and any treatment targeting tumor immune pathway
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplantation
* Positive test for human immunodeficiency virus,Active hepatitis B or hepatitis C
* Receipt of a live, attenuated vaccine within 30 days prior to randomization, during treatment
* Pregnancy or lactation
* Dysphagia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2028-08-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rates (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1
Number of participants with adverse events (AEs) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  Disease control rate (DCR) is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST V1.1
Duration of response (DOR) | Up to approximately 2 years
  DOR is defined for participants who had an objective response as the time from the first occurrence of a documented confirmed response (CR or PR) to the date of disease progression per RECIST v1.1 or death from any cause,whichever occurred first
Time to response (TTR) | Up to approximately 2 years
  TTR is defined for participants who had an objective response as the time from the start of treatment to the first occurrence of a documented unconfirmed response (CR or PR) .
Progression-free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the start of treatment till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Progression-free survival 2 (PFS2) | Up to approximately 2 years
  PFS 2 is defined as the time from the start of treatment till the second documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Overall survival (OS) | Up to approximately 2 years
  Overall survival is defined as the time from the start of treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Summit Therapeutics Research Site, Los Angeles, California
  - Summit Therapeutics Research Site, Murrieta, California
  - Summit Therapeutics Research Site, Fairfax, Virginia
- The Sixth Hospital,Sun Yat-sen University, Guanzhou, Guangdong, China